CLINICAL TRIAL: NCT04660292
Title: Clinical Outcomes of Maitland's Mobilization in Patients With Myofacial Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Maryam Shabbir, Associate Professor, Riphah International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT-Associate-MARYAM SHABBIR
Record Dates: First submitted 2020-12-01; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Myofascial Pain Syndrome of Neck
Keywords: Neck Pain; Manual mobilization; Isometric exercise; Triger points; Visual analog scale
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): The study group was treated with Maitland mobilization and manipulation techniques including postero-anterior Maitland mobilization for C1-C2, Maitland lateral PA glide for C3-C6 and Maitland thrust manipulation for cervico-thoracic junction. Frequency of mobilization was 2 days a week for 4 weeks. While intensity of mobilization was grade 3 and 4 based on the Maitland concept.13 Time of oscillations was 2 or 3 oscillations in a second for 1 to 2 minutes.
  Interventions: Other: Maitland's mobilization
- Control Group (Active Comparator): While placebo treatment with conventional physiotherapy (active exercises-10 repetitions in all direction in pain free range, isometrics 5-10 seconds brief but maximum contraction each held for 5-16 seconds for flexors, extensors, side flexors and rotators)14 without gliding, oscillations and thrust were recommended for the control group.The placebo group was treated with baseline treatment including TENS 10 minutes and moist hot packs in sitting position for 15 minutes on cervical region in with head resting on table with a pillow.
  Interventions: Other: Traditional Physical therapy

INTERVENTIONS:
Other: Maitland's mobilization — Maitland's techniques involve the application of passive and accessory oscillatory movements to spinal and vertebral joints to treat pain and stiffness.It has Five grades
  Arms: Study Group
Other: Traditional Physical therapy — BASELINE TREATMENT INCLUDES TENS and Hot PACKS
  Arms: Control Group

SUMMARY:
Myofacial neck pain is a common musculoskeletal problem caused by presence of trigger points and local and referred pain patterns. Chronic neck pain is responsible for the involvement of joints, ligaments, fascia and connective tissue as well. The objective of this study was to assess the impacts of Maitland's mobilization in patients with myofacial chronic neck pain. Maitland's mobilization is one of the most common manual therapy approaches used by physiotherapists. Maitland's techniques involve the application of passive and accessory oscillatory movements to spinal and vertebral joints to treat pain and stiffness.

In this randomized, placebo treatment controlled trial, 30 patients consecutively aged 25-45 years meeting inclusion criteria were isolated into two groups. The study group was treated with Maitland's mobilization consistently for 8 weeks while the control group got placebo treatment for a similar time frame. Visual analog Scale (VAS), Neck disability index (NDI) and cervical range of motion (ROM) questionnaire was filled by patients before, intermediate and after the intervention to evaluate the severity of pain, functional ability and range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 25-45 years old,
* Bilateral pain involving the upper trapezius and elevator muscle of the scapula;
* Duration of pain of at least 3 months;
* A pain intensity corresponding to at least 2 cm on a 10 cm visual analogue scale (VAS); -Neck pain with symptoms provoked by either neck postures or neck movement;
* Pain localized at least in the cervical and occipital regions but not in the orofacial region; --Neck disability index (NDI) greater than or equal to 15 points;
* Restricted cervical range of movements (flexion, extension, rotation, and side-bending); ---Presence of bilateral MTrPs in upper trapezius and levator scapulae muscles were included in this study.

Exclusion Criteria:

* A history of traumatic injuries (e.g., contusion, fracture, and whiplash injury);
* Systemic diseases such as fibromyalgia, systemic erythematous lupus and arthritis;
* Neurologic disorders (e.g., trigeminal neuralgia or occipital neuralgia);
* Concomitant medical diagnosis of any primary headache (tension type or migraine);
* Cervical spine surgery; and clinical diagnosis of cervical radiculopathy or myelopathy

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 2 months
  Its a pain rating Scale Scoring between 0-10.O means no pain 10 means worse pain
Neck disability Index | 2 months
  Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Shabbir, PhD*, Principal Investigator — Riphah International University; Naveed Arshad, Mphil, Principal Investigator — Islamabad Medical and Dental College
Locations (1):
- Riphah IU, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsieh YL, Kao MJ, Kuan TS, Chen SM, Chen JT, Hong CZ. Dry needling to a key myofascial trigger point may reduce the irritability of satellite MTrPs. Am J Phys Med Rehabil. 2007 May;86(5):397-403. doi: 10.1097/PHM.0b013e31804a554d. PMID 17449984
- [Background] Leon-Hernandez JV, Martin-Pintado-Zugasti A, Frutos LG, Alguacil-Diego IM, de la Llave-Rincon AI, Fernandez-Carnero J. Immediate and short-term effects of the combination of dry needling and percutaneous TENS on post-needling soreness in patients with chronic myofascial neck pain. Braz J Phys Ther. 2016 Jul 11;20(5):422-431. doi: 10.1590/bjpt-rbf.2014.0176. PMID 27410163
- [Background] Gattie E, Cleland JA, Snodgrass S. The Effectiveness of Trigger Point Dry Needling for Musculoskeletal Conditions by Physical Therapists: A Systematic Review and Meta-analysis. J Orthop Sports Phys Ther. 2017 Mar;47(3):133-149. doi: 10.2519/jospt.2017.7096. Epub 2017 Feb 3. PMID 28158962
- [Background] Tekin L, Akarsu S, Durmus O, Cakar E, Dincer U, Kiralp MZ. The effect of dry needling in the treatment of myofascial pain syndrome: a randomized double-blinded placebo-controlled trial. Clin Rheumatol. 2013 Mar;32(3):309-15. doi: 10.1007/s10067-012-2112-3. Epub 2012 Nov 9. PMID 23138883
- [Background] Yeganeh Lari A, Okhovatian F, Naimi Ss, Baghban AA. The effect of the combination of dry needling and MET on latent trigger point upper trapezius in females. Man Ther. 2016 Feb;21:204-9. doi: 10.1016/j.math.2015.08.004. Epub 2015 Aug 14. PMID 26304789
- [Background] Clewley D, Flynn TW, Koppenhaver S. Trigger point dry needling as an adjunct treatment for a patient with adhesive capsulitis of the shoulder. J Orthop Sports Phys Ther. 2014 Feb;44(2):92-101. doi: 10.2519/jospt.2014.4915. Epub 2013 Nov 21. PMID 24261931
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405